CLINICAL TRIAL: NCT04197687
Title: Phase II Trial to Evaluate Immune-Related Biomarkers for Pathological Response in Stage II-III HER2-Positive Breast Cancer Receiving Neoadjuvant Chemotherapy With Subsequent Randomization to Multi-Epitope HER2 Vaccine vs. Placebo in Patients With Residual Disease Post-Neoadjuvant Chemotherapy
Brief Title: TPIV100 and Sargramostim for the Treatment of HER2 Positive, Stage II-III Breast Cancer in Patients With Residual Disease After Chemotherapy and Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC1835-ACCRU-BR-1701; NCI-2019-08038 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1835-ACCRU-BR-1701 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2019-12-05; First posted 2019-12-13 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-05

CONDITIONS: Breast Adenocarcinoma; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; 2C4 antibody; sargramostim; Colony-Stimulating Factors; Trastuzumab; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I - No pCR (trastuzumab emtansine, TPIV100, sargramostim) (Experimental): Patients receive standard of care maintenance therapy with trastuzumab emtansine and receive TPIV100 ID and sargramostim ID on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive two additional booster injections of TPIV100 ID and sargramostim ID at 3 and 12 months after completion of trastuzumab emtansine maintenance therapy.
  Interventions: Biological: Multi-epitope HER2 Peptide Vaccine TPIV100; Biological: Sargramostim; Biological: Trastuzumab Emtansine
- Arm II - No pCR (trastuzumab emtansine, placebo, sargramostim) (Placebo Comparator): Patients receive standard of care maintenance therapy with trastuzumab emtansine and receive placebo ID and sargramostim ID on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive two additional booster injections of placebo ID and sargramostim ID at 3 and 12 months after completion of trastuzumab emtansine maintenance therapy.
  Interventions: Other: Placebo Administration; Biological: Sargramostim; Biological: Trastuzumab Emtansine
- Treatment (pCR) (Experimental): Patients receive standard of care maintenance therapy with trastuzumab and pertuzumab for 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pertuzumab; Biological: Trastuzumab

INTERVENTIONS:
Biological: Multi-epitope HER2 Peptide Vaccine TPIV100 — Given ID
  Other Names: HER2/Neu Peptide Vaccine TPIV100; Peptide Vaccine TPIV100; TPIV 100; TPIV-100; TPIV100
  Arms: Arm I - No pCR (trastuzumab emtansine, TPIV100, sargramostim)
Biological: Pertuzumab — permitted at physician's discretion
  Other Names: 2C4; 2C4 Antibody; HS627; MoAb 2C4; Monoclonal Antibody 2C4; Omnitarg; Perjeta; Pertuzumab Biosimilar HS627; rhuMAb2C4; RO4368451
  Arms: Treatment (pCR)
Other: Placebo Administration — Given ID
  Arms: Arm II - No pCR (trastuzumab emtansine, placebo, sargramostim)
Biological: Sargramostim — Given ID
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
  Arms: Arm I - No pCR (trastuzumab emtansine, TPIV100, sargramostim); Arm II - No pCR (trastuzumab emtansine, placebo, sargramostim)
Biological: Trastuzumab — therapy are at the discretion of the treating physicians
  Other Names: ABP 980; ALT02; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herzuma; Kanjinti; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; Ontruzant; PF-05280014; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-pkrb; Trastuzumab-qyyp; Trazimera
  Arms: Treatment (pCR)
Biological: Trastuzumab Emtansine — at the discretion of the treating physicians.
  Other Names: Ado Trastuzumab Emtansine; ADO-Trastuzumab Emtansine; Kadcyla; PRO132365; RO5304020; T-DM1; Trastuzumab-DM1; Trastuzumab-MCC-DM1; Trastuzumab-MCC-DM1 Antibody-Drug Conjugate; Trastuzumab-MCC-DM1 Immunoconjugate
  Arms: Arm I - No pCR (trastuzumab emtansine, TPIV100, sargramostim); Arm II - No pCR (trastuzumab emtansine, placebo, sargramostim)

SUMMARY:
This phase II trial studies how well TPIV100 and sargramostim work in treating patients with HER2 positive, stage II-III breast cancer that has residual disease after chemotherapy prior to surgery. It also studies why some HER2 positive breast cancer patients respond better to chemotherapy in combination with trastuzumab and pertuzumab. TPIV100 is a type of vaccine made from HER2 peptide that may help the body build an effective immune response to kill tumor cells that express HER2. Sargramostim increases the number of white blood cells in the body following chemotherapy for certain types of cancer and is used to alert the immune system. It is not yet known if TPIV100 and sargramostim will work better in treating patients with HER2 positive, stage II-III breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate invasive disease free survival (iDFS) of multi-epitope HER2 vaccine versus (vs.) placebo in combination with ado-trastuzumab emtansine (TTT-DM1) in patients with stage II-III HER2 positive (+) breast cancer (BC) with residual disease post-neoadjuvant chemotherapy.

II. To evaluate the safety of multi-epitope HER2 vaccine given concurrently with ado-trastuzumab emtansine (T-DM1) maintenance therapy.

SECONDARY OBJECTIVES:

I. To evaluate immunogenicity of multi-epitope HER2 vaccine in combination with T-DM1 maintenance therapy.

II. To evaluate the immune-related tissue and blood biomarkers for complete pathological response in patients with stage II-III HER2+ BC receiving neoadjuvant chemotherapy.

CORRELATIVE RESEARCH OBJECTIVES:

I. To determine host immune factors which are critical to prevent disease recurrence in HER2+ BC patients.

Ia. To determine if the development of T cell immunity, as assessed by IFN-gamma enzyme-linked immunospot (ELISpot), to HER2 correlates with improved iDFS.

Ib. To determine the distribution of the helper T cell response among helper T cell differentiation states.

Ic. To determine if augmenting CD4 helper T cell immunity augments HER2-specific antibody immunity induced by trastuzumab.

Id. To determine if human leukocyte antigen (HLA) genotypes are associated with antibody responses before and after neoadjuvant therapy and vaccination.

Ie. To determine gene expression levels in tumors from patients who did not achieve complete pathological response (pCR) that are associated with recurrence.

II. To determine tumor intrinsic genotyping and phenotyping features associated with therapeutic failure to HER2 immune-based approaches.

IIa. To determine whether HER2 monoclonal antibody therapy induces HER2 loss and modulation of HER2-specific adaptive immune responses.

IIb. To determine loss-of-function mutations in breast tumor that associate with lack of pCR and lack of immune response to HER2+ neoadjuvant treatment.

OUTLINE:

pCR AFTER NEOADJUVANT CHEMOTHERAPY AND SURGERY: Patients receive standard of care maintenance therapy with trastuzumab and pertuzumab for 1 year in the absence of disease progression or unacceptable toxicity.

NO pCR AFTER NEOADJUVANT CHEMOTHERAPY AND SURGERY: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care maintenance therapy with trastuzumab emtansine and receive TPIV100 intradermally (ID) and sargramostim ID on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive two additional booster injections of TPIV100 ID and sargramostim ID at 3 and 12 months after completion of trastuzumab emtansine maintenance therapy.

ARM 2: Patients receive standard of care maintenance therapy with trastuzumab emtansine and receive placebo intradermally (ID) and sargramostim ID on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive two additional booster injections of placebo ID and sargramostim ID at 3 and 12 months after completion of trastuzumab emtansine maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Histologically confirmed adenocarcinoma of the breast stage >= T2 OR >= N1 based on the 7th edition of tumor, node, metastases (TNM) staging system from the American Joint Committee on Cancer
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Any estrogen receptor (ER) or progesterone receptor (PR) but HER2 positive defined as 3+ staining intensity (on a scale of 0 to 3) by means of immunohistochemistry (IHC) analysis OR gene amplification on fluorescence in situ hybridization (FISH) ratio >= 2.0
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Willingness to provide adequate pretreatment biopsy sample

  * NOTE: Adequate tissue samples defined as core needle biopsy or incisional biopsy or excisional samples that can provide >= 3 core needle biopsies with at least 14 gauge (G) needle with 12 unstained sections of 5 micron thickness. Fine needle aspiration (FNA) sample alone is not sufficient
  * NOTE: Patients without adequate pretreatment biopsy samples must be agreeable to have an additional research biopsy prior to neoadjuvant therapy
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, 2
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Willing to employ adequate contraception from the time of pre-registration through 6 months after the final vaccine cycle
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Willing to receive a tetanus vaccination if subject has not had one =< 1 year prior to pre-registration
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Provide written informed consent
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Willing to provide mandatory tissue and blood samples for correlative research purposes
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Negative pregnancy test done =< 7 days prior to pre-registration, for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* REGISTRATION (SAFETY LEAD-IN): Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 28 days prior to registration)
* REGISTRATION (SAFETY LEAD-IN): Platelet count >= 75,000/mm^3 (obtained =< 28 days prior to registration)
* REGISTRATION (SAFETY LEAD-IN): Hemoglobin >= 9.0 g/dL (obtained =< 28 days prior to registration)
* REGISTRATION (SAFETY LEAD-IN): Direct bilirubin < 1.5 x upper limit of normal (ULN) (obtained =< 28 days prior to registration)
* REGISTRATION (SAFETY LEAD-IN): Aspartate transaminase (AST) =< 3 x ULN (obtained =< 28 days prior to registration)
* REGISTRATION (SAFETY LEAD-IN): Creatinine =< 2 x ULN (obtained =< 28 days prior to registration)
* REGISTRATION (SAFETY LEAD-IN): Prothrombin time (PT)/international normalized ratio (INR)/ partial thromboplastin time (PTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and PT or PTT is within therapeutic range of intended use of coagulant (obtained =< 28 days prior to registration)
* REGISTRATION (SAFETY LEAD-IN): Completed planned curative breast surgeries (not including any future breast reconstructive surgery) and any radiation therapy >= 30 days prior to registration
* REGISTRATION (SAFETY LEAD-IN): Completed last cycle of chemotherapy >= 90 days prior to registration

  * NOTE: Prior to registration, patients must not receive > 8 cycles of TDM-1 maintenance therapy after surgery
* REGISTRATION (SAFETY LEAD-IN): Any residual disease after trastuzumab +/- pertuzumab based neoadjuvant chemotherapy warranted T-DM1 as per treating physician
* REGISTRATION (SAFETY LEAD-IN): Adequate tissue specimens from both pre-treatment biopsy and surgery must be submitted. Adequate tissue samples defined as core needle biopsy or incisional biopsy or excisional samples that can provide >= 3 core needle biopsies with at least 14G needle with 12 unstained sections of 5 micron thickness

  * NOTE: Fine needle aspiration (FNA) sample alone is not sufficient
* REGISTRATION (SAFETY LEAD-IN): Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* REGISTRATION (SAFETY LEAD-IN): ECOG performance status (PS) 0, 1, 2
* REGISTRATION (SAFETY LEAD-IN): Willing to employ adequate contraception from the time of registration through 6 months after the final vaccine cycle
* REGISTRATION - FOR PATIENTS WITH NO RESIDUAL DISEASE (pCR) - (PHASE II): ECOG performance status (PS) 0, 1, 2
* REGISTRATION - FOR PATIENTS WITH NO RESIDUAL DISEASE (pCR) - (PHASE II): Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 28 days prior to registration)
* REGISTRATION - FOR PATIENTS WITH NO RESIDUAL DISEASE (pCR) - (PHASE II): Platelet count >= 75,000/mm^3 (obtained =< 28 days prior to registration)
* REGISTRATION - FOR PATIENTS WITH NO RESIDUAL DISEASE (pCR) - (PHASE II): Hemoglobin >= 9.0 g/dL (obtained =< 28 days prior to registration)
* REGISTRATION - FOR PATIENTS WITH NO RESIDUAL DISEASE (pCR) - (PHASE II): Direct bilirubin < 1.5 x upper limit of normal (ULN) (obtained =< 28 days prior to registration)
* REGISTRATION - FOR PATIENTS WITH NO RESIDUAL DISEASE (pCR) - (PHASE II): Aspartate transaminase (AST) =< 3 x ULN (obtained =< 28 days prior to registration)
* REGISTRATION - FOR PATIENTS WITH NO RESIDUAL DISEASE (pCR) - (PHASE II): Calculated serum creatinine clearance of >= 50 mL/minute (min.) (obtained =< 28 days prior to registration)
* REGISTRATION - FOR PATIENTS WITH NO RESIDUAL DISEASE (pCR) - (PHASE II): PT/INR/PTT =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and PT or PTT is within therapeutic range of intended use of coagulants (obtained =< 28 days prior to registration)
* REGISTRATION - FOR PATIENTS WITH NO RESIDUAL DISEASE (pCR) - (PHASE II): Negative pregnancy test done =< 7 days prior to registration, for person of childbearing potential

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 28 days prior to randomization)
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): Platelet count >= 75,000/mm^3 (obtained =< 28 days prior to randomization)
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): Hemoglobin >= 9.0 g/dL (obtained =< 28 days prior to randomization)
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): Direct bilirubin < 1.5 x upper limit of normal (ULN) (obtained =< 28 days prior to randomization)
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): Aspartate transaminase (AST) =< 3 x ULN (obtained =< 28 days prior to randomization)
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): Creatinine =< 2 x ULN (obtained =< 28 days prior to randomization)
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): PT/INR/PTT =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and PT or PTT is within therapeutic range of intended use of coagulant (obtained =< 28 days prior to randomization)
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): Completed last cycle of chemotherapy >= 90 days prior to randomization

  * NOTE: Prior to randomization, patients must not receive >= 6 cycles of T-DM1 maintenance therapy after surgery
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): Have residual disease with >= 1 cm residual tumor in the breast (>= ypT1c) and/or persistent lymph node positivity after trastuzumab +/- pertuzumab based neoadjuvant chemotherapy
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): Adequate tissue specimens from both pre-treatment biopsy and surgery must be submitted. Adequate tissue samples defined as core needle biopsy or incisional biopsy or excisional samples that can provide >= 3 core needle biopsies with at least 14G needle with 12 unstained sections of 5 micron thickness

  * NOTE: Fine needle aspiration (FNA) sample alone is not sufficient
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): Negative pregnancy test done =< 7 days prior to randomization, for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): ECOG performance status (PS) 0, 1, 2
* RANDOMIZATION - PATIENTS WITH RESIDUAL DISEASE POST NEOADJUVANT TRATUZUMAB +/- PERTUZUMAB BASED CHEMOTHERAPY (NO pCR) - (PHASE II): Willing to employ adequate contraception from the time of randomization through 6 months after the final vaccine cycle

Exclusion Criteria:

* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant person
  * Nursing person unwilling to stop breast feeding
  * Person of child bearing potential who are unwilling to employ adequate contraception from the time of registration through 6 months after the final vaccine cycle
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Clinical evidence of active local recurrence or distant metastases

  * NOTE: All patients must have either a positron emission tomography (PET)/computed tomography (CT) or CT chest, abdomen, and pelvis with bone scan to rule out distant metastases =< 365 days prior to preregistration. If any of these is concerning, follow-up imaging or biopsy should be performed if indicated rule out distant metastases
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Immunocompromised patients including patients known to be human immunodeficiency virus (HIV) positive or those on chronic steroids

  * NOTE: Must be off systemic steroids at least 14 days prior to pre-registration. However, topical steroids, inhalants or steroid eye drops are permitted
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Uncontrolled acute or chronic medical conditions including, but not limited to the following:

  * Active infection requiring antibiotics
  * Congestive heart failure with New York Heart Association class III or IV; moderate to severe objective evidence of cardiovascular disease
  * Myocardial infarction or stroke =< 6 months prior to pre-registration
  * Significant cardiac arrhythmia or unstable angina
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Receiving any other investigational agent
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Other active malignancy at time of pre-registration or =< 3 years prior to preregistration

  * EXCEPTIONS: Non-melanoma skin cancer or carcinoma-in-situ (e.g. of cervix, prostate)
  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment (cytotoxics, monoclonal antibodies, small molecule inhibitors) for their cancer
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Known history of active autoimmune disease that has required systemic treatment in the =< 30 days (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) prior to pre-registration. NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Patients with vitiligo, Graves disease, or psoriasis not requiring systemic treatment within the past 30 days are not excluded. Patients with Celiac disease controlled with diet modification are not excluded
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Any prior hypersensitivity or adverse reaction to granulocyte-macrophage colony stimulating factor (GM-CSF)
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): History of trastuzumab-related cardiac toxicity requiring interruption or discontinuation of therapy, even if left ventricular ejection fraction (LVEF) fully recovered
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Baseline LVEF < 50%
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): History of myocardial infarction =< 168 days (6 months) prior to pre-registration, or congestive heart failure requiring use of ongoing maintenance therapy for life threatening ventricular arrhythmias
* PRE-REGISTRATION FOR ALL PATIENTS (INCLUDE SAFETY LEAD-IN): Patients who received tamoxifen or raloxifene or another agent for prevention of breast cancer =< 2 months prior to pre-registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (iDFS) between the 2 arms | From time of randomization to recurrence, invasive breast cancer or death, assessed up to 5 years
  iDFS will be defined from the time of randomization to ipsilateral invasive breast tumor recurrence, regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause, contralateral invasive breast cancer, or second primary non-breast invasive cancer. Will be based on stratified log-rank test at one-sided 0.01 level in an intention-to-treat population, where the stratification is by the randomization stratification factors. The Cox proportional hazards model will be used to adjust for the trial stratification factors (hormone receptor, human leukocyte antigen A classification, status and clinical stage). Subgroup analyses of iDFS will also be performed by stratification factors and other baseline characteristics, with the caveat that statistical power for these subgroup analyses may be limited.

SECONDARY OUTCOMES:
Overall survival | From randomization to the date of death due to any cause, assessed up to 5 years
  defined as the time from randomization to the date of death due to any cause. Patients who are lost to follow-up for OS will be censored at the date the subject was last known to be alive
Incidence of adverse events (AEs) | Up to 24 months
  Will be assessed according to Common Terminology Criteria for Adverse Events 5.0 and defined as adverse events that are classified as either unrelated, unlikely to be related, possibly, probably, or definitely related to the study treatment. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed by primary disease site to determine toxicity patterns. Frequency tables will be generated to summarize the occurrence of treatment-related AE's by treatment arms. Comparisons of the rates of individual AE's will be done using tests of proportions such as Fisher's exact test or Chi-squared test. Additional analysis will use the Cochran-Mantel-Haenszel chi-squared test with study stratification factors.
Immunogenicity assessment | Up to 5 years
  To evaluate immunogenicity of multi-epitope HER2 vaccine in combination with T-DM1 maintenance therapy.
Complete pathological response | Baseline
  Will be assessed using immune-related tissue and blood biomarkers.
Vaccine induced HER2-specific T cell responses | Baseline up to 24 months
  Will be defined as a 2-fold or greater increase in HER2-specific antibody concentration from pre-treatment levels at any point during treatment or HER2-specific antibodies above the lower limit of detection at any point during treatment if pre-treatment levels were non-detectable. Antibody response frequency at the post-treatment initiation time points will be compared among arms using a chi-squared test. Antibody response magnitude at the post-treatment initiation time point will be compared among arms using an analysis of variance F-test followed by Tukey pairwise comparisons between pairs of arms. Likelihood of antibody response at the post-treatment initiation time point will be compared among arms using logistic regression (the dependent variable is antibody response [yes/no] at the post-treatment initiation time point; the independent variables are the antibody response [yes/no] at the pre-treatment time point and a categorical variable capturing arm).

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, Principal Investigator — Mayo Clinic
Locations (30):
- United States (30):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Middlesex Hospital, Middletown, Connecticut
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Cleveland Clinic Florida, West Palm Beach, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Carle Cancer Center NCI Community Oncology Research Program, Urbana, Illinois
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - University Medical Center New Orleans, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Essentia Health NCI Community Oncology Research Program, Duluth, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Lexington Medical Center, West Columbia, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin